CLINICAL TRIAL: NCT01386554
Title: A Randomized, Placebo-Controlled, Parallel-Group, Double-Blind Study of H.P. Acthar Gel (Acthar) in Treatment-Resistant Subjects With Persistent Proteinuria and Nephrotic Syndrome Due to Idiopathic Membranous Nephropathy (iMN)
Brief Title: Acthar for Treatment of Proteinuria in Membranous Nephropathy Patients
Acronym: CHART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QSC01-MN-01; Control No. 166679 (Other: Health Canada)
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2018-04

CONDITIONS: Proteinuria; Idiopathic Membranous Nephropathy
Keywords: H.P. Acthar Gel; Acthar; nephrotic syndrome; idiopathic membranous nephropathy; proteinuria
MeSH Terms: conditions — Proteinuria; Glomerulonephritis, Membranous; Nephrotic Syndrome | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 80 U Acthar (Experimental): Acthar (Repository Corticotropin Injection) 80 U (1.0 mL) two times per week
  Interventions: Drug: Repository Corticotropin Injection
- 1.0 mL Placebo (Placebo Comparator): Placebo (1.0 mL) two times per week
  Interventions: Drug: Placebo
- 40 U Acthar (Experimental): Acthar (Repository Corticotropin Injection) 40 U (1.0 mL) two times per week
  Interventions: Drug: Repository Corticotropin Injection

INTERVENTIONS:
Drug: Repository Corticotropin Injection — Acthar given SC for 6 months
  Other Names: H.P. Acthar Gel; ACTH Gel; ACTH
  Arms: 40 U Acthar; 80 U Acthar
Drug: Placebo — Placebo contains the same inactive ingredients as that used for H.P. Acthar Gel without the API.
  Placebo given SC for 6 months (80 U two times a week).
  Arms: 1.0 mL Placebo

SUMMARY:
The purpose of this study is to provide nephrologists with additional clinical evidence regarding the efficacy and safety of Acthar in subjects with treatment-resistant idiopathic membranous nephropathy. Approximately sixty (60) subjects will be randomized in this double-blind, parallel-group, placebo-controlled, multicenter study comparing Acthar and Placebo administered 2 times per week for a 24-week treatment period followed by a 24-week observation period. The primary objective of this study is to assess the proportion of treatment-resistant subjects (defined as subjects who either have had no response or have suffered a relapse after achieving a partial response to their most recent standard treatment regimen) who have a complete or partial remission of proteinuria in nephrotic syndrome due to idiopathic membranous nephropathy after 24 weeks of treatment.

ELIGIBILITY:
For complete list of inclusion and exclusion criteria, please refer to contact below.

Inclusion Criteria:

* Male or female subjects ≥18 years of age, at screening Visit 1:

  a. If potential subjects are >75 years of age, discussion between the investigator and the Medical Monitor must take place;
* Body mass index ≤40 kg/m2, at screening Visit 1;
* A history of nephrotic syndrome due to iMN as confirmed by documented results from a renal biopsy performed within 4 years prior to screening Visit 1:

  a. If a biopsy has been performed between 4-8 years prior to screening, and if the subject has no signs or symptoms of diabetes or other clinical diagnoses that could suggest a change in renal histology in the opinion of the investigator and the Medical Monitor, the subject is eligible.
* Renal target disease requirements:

  1. Total urine protein of ≥3.0g (≥3000mg) from the 24-hour urine returned at Visit 1A, AND.
  2. An estimated glomerular filtration rate (eGFR) value >25mL/min/1.73m2 at Visit 1A (as calculated using the abbreviated Modification of Diet in Renal Disease [MDRD] equation.
* Any prior course of at least 1 month of treatment with ≥1 of an immunosuppressant therapy(ies) for iMN:

  1. Subjects must be followed for at least 3 months after treatment prior to screening with the exception of rituximab or a cytotoxic based therapy, where the follow-up period is 6 months after treatment. If after follow-up it was determined that the subject did not achieve a complete or partial remission or suffered a relapse after achieving a partial remission, the subject will be eligible for the study.
  2. If in the investigator's opinion, the subject should be enrolled prior to meeting the follow-up period criteria and the decrease in proteinuria is no longer occurring, discussion between the investigator and the Medical Monitor must take place for approval to enter screening.
* History of treatment-resistant iMN defined as either having had no remission or having suffered a relapse after achieving a partial remission to their most recent standard treatment regimen as defined in the Definition of Response Status Table despite treatment with at least 1 month of treatment with a prior therapy for iMN. Note the following:

  a. If the subject has been treated with prior standard therapy and can no longer be re-treated with any component of that therapy, regardless of whether a complete or partial remission was achieved, then the subject may be eligible, but approval from the Medical Monitor is required.

  i. For example, if early discontinuation of standard therapy occurred because of a serious adverse event (Grade 3 or 4) during the treatment, regardless of whether a partial or complete remission was achieved, then the subject may be eligible.

  b. If (a) does not apply, and the subject did not have either a partial or complete remission to the most recent treatment regimen, then the subject is eligible.

  c. If (a) does not apply, and the subject achieved a partial remission from the most recent treatment regimen, and later relapse occurred, then the subject is eligible.
* Antihypertensive treatment including use of ACE inhibitors and/or ARB:

  a. Unless there is a history of intolerance to ACE inhibitors or ARB therapy, the subject must be treated with at least one of these agents.

  b. Treatment with ACE inhibitor and/or ARB for ≥3 months prior to screening Visit 1A, with stable maintenance dose for ≥30 days prior to randomization.

  c. If treated with other antihypertensive therapies, treatment duration of ≥30 days and stable maintenance dose for ≥7 days prior to screening Visit 1A.
* Blood pressure determined by the average of ≥3 seated readings taken ≥5 minutes apart during the screening period at Visit 1A:

  1. Mean systolic blood pressure ≤140 mmHg and
  2. Mean diastolic blood pressure ≤80 mmHg.

Exclusion Criteria:

* Therapies and/or medications:

  1. History of previous use of Acthar for treatment of nephrotic syndrome;
  2. Prior sensitivity to Acthar or other porcine protein products; or
  3. Planned treatment with live or live attenuated vaccines once enrolled in the study.
* Contraindication to Acthar per Prescribing Information: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenocortical hyperfunction.

  a. For the purpose of this study: "history" of peptic ulcer is defined as ≤6 months prior to Visit 1A.
* Renal target disease exclusions:

  1. Subjects with known diabetic nephropathy or nephrotic syndrome due to a disease or process other than idiopathic membranous nephropathy, or
  2. Subjects requiring diagnostic or interventional procedure requiring a contrast agent must delay screening/randomization for at least 7 days.
* History of Systemic Lupus Erythematosus.
* Type 1 or Type 2 diabetes mellitus (prior diagnosis of gestational diabetes mellitus is not an exclusion).
* History of Deep Vein Thrombosis (DVT) ≤6 months prior to screening Visit 1A.
* Presence of renal vein thrombosis:

  1. Known current diagnosis by ultrasound, magnetic resonance imaging (MRI) or computed tomography scan;
  2. Signs or symptoms consistent with occurrence of acute renal vein thrombosis (hematuria in combination with flank pain and >30% unexplained acute rise in serum creatinine) with renal vein thrombosis confirmed by ultrasound, MRI or computed tomography scan.
* Cardiovascular exclusions:

  1. History of or active congestive heart failure (NYHA Functional Classification of CHF Class II through Class IV), or.
  2. History of known dilated cardiomyopathy with left ventricular ejection fraction ≤40%, or.
  3. Occurrence of any of the following within 3 months of screening Visit 1A:

  i. Unstable angina. ii. Myocardial infarction. iii. Coronary artery bypass graft or percutaneous transluminal coronary angioplasty.

iv. Transient ischemic attack or cerebrovascular disease. v. unstable arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2016-11-21 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (28):
- United States (14):
  - Mallinckrodt Investigational Site, Sacramento, California
  - Mallinckrodt Investigational Site, Stanford, California
  - Mallinckrodt Investigational Site, Jacksonville, Florida
  - Mallinckrodt Investigational Site, Atlanta, Georgia
  - Mallinckrodt Investigational Site, Rochester, Minnesota
  - Mallinckrodt Investigational Site, Reno, Nevada
  - Mallinckrodt Investigational Site, New York, New York
  - Mallinckrodt Investigational Site, Chapel Hill, North Carolina
  - Mallinckrodt Investigational Site, Durham, North Carolina
  - Mallinckrodt Investigational Site, Bethlehem, Pennsylvania
  - Mallinckrodt Investigational Site, Charleston, South Carolina
  - Mallinckrodt Investigational Site, Chattanooga, Tennessee
  - Mallinckrodt Investigational Site, Houston, Texas
  - Mallinckrodt Investigational Site, Lubbock, Texas
- Mallinckrodt Investigational Site, Toronto, Ontario, Canada
- Chile (2):
  - Mallinckrodt Investigational Site, La Serena, Coquimbo Region
  - Mallinckrodt Investigational Site, Temuco
- Mexico (2):
  - Mallinckrodt Investigational Site, Monterrey, Nuevo León
  - Mallinckrodt Investigational Site, San Nicolás de los Garza, Nuevo León
- Turkey (Türkiye) (9):
  - Mallinckrodt Investigational Site 307, Adana
  - Mallinckrodt Investigational Site 305, Ankara
  - Mallinckrodt Investigational Site 308, Ankara
  - Mallinckrodt Investigational Site 302, Antalya
  - Mallinckrodt Investigational Site 301, Istanbul
  - Mallinckrodt Investigational Site 309, Istanbul
  - Mallinckrodt Investigational Site 303, Izmir
  - Mallinckrodt Investigational Site 310, Kocaeli
  - Mallinckrodt Investigational Site 304, Mersin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bomback AS, Tumlin JA, Baranski J, Bourdeau JE, Besarab A, Appel AS, Radhakrishnan J, Appel GB. Treatment of nephrotic syndrome with adrenocorticotropic hormone (ACTH) gel. Drug Des Devel Ther. 2011 Mar 14;5:147-53. doi: 10.2147/DDDT.S17521. PMID 21448451
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United Staes. The first participant was screened on 20 October 2011. The last study visit occurred on 05 May 2017.
Pre-assignment Details: 132 participants were screened.
Groups:
- Acthar 40U: 40 units (U) of Acthar administered 5 times a week
- Acthar 80U: 80 U of Acthar administered 2 times a week
- Combined Placebo: Placebo (volume matched for 40 U or 80 U) administered 5 times (40 U) or 2 times (80 U) per week
Period: Overall Study
Arm/Group | Acthar 40U | Acthar 80U | Combined Placebo
Started | 4 | 35 | 21
Completed | 1 | 26 | 15
Not Completed | 3 | 9 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 2 | 5 | 2
Not completed — Progressive disease | 1 | 2 | 2
Not completed — Administration of live vaccines | 0 | 1 | 0
Not completed — Investigator discretion | 0 | 0 | 1
Not completed — Reason not collected | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received ≥ 1 dose of study medication.
Groups:
- Acthar 40U: 40 U of Acthar administered 5 times a week
- Combined Placbeo: Placebo (volume matched for 40 U or 80 U) administered 5 times (40 U) or 2 times (80 U) per week
- Total: Total of all reporting groups
Arm/Group | Acthar 40U | Acthar 80U | Combined Placbeo | Total
Number analyzed (Participants) | 4 | 35 | 21 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (5.72) | 49.9 (13.18) | 45.4 (12.24) | 48.7 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 4 | 15
  Male | 2 | 26 | 17 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 1 | 0 | 2
  Turkey | 0 | 6 | 4 | 10
  United States | 3 | 15 | 10 | 28
  Mexico | 0 | 4 | 1 | 5
  Chile | 0 | 3 | 2 | 5
  Argentina | 0 | 6 | 2 | 8
  Colombia | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete or Partial Remission in Proteinuria at 24 Weeks
Description: The participant's response was considered the average of the two PCR values from the 24-hour urine collected at Visit 8 (Week 24). Urine protein creatinine ratio (uPCR) was used to assess remission (partial and complete). Complete remission = uPCR < 0.3 g/g; partial remission = uPCR < 50% of baseline uPCR and > 0.3 g/g but < 3.0 g/g.
Time Frame: At Visit 8 (Week 24)
Population: ITT Population included all randomized participants who received ≥ 1 dose of study mediation and who contributed any efficacy data in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar 40U | Acthar 80U | Combined Placebo
Number analyzed (Participants) | 4 | 35 | 21
Participants
  Partial remission in proteinuria | 1 | 5 | 2
  Complete remission in proteinuria | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With Sustained Remission
Description: The participant's response was considered the average of the two PCR values from the 24-hour urine collections at Visit 8 (Week 24).
Time Frame: At Visit 9 (Week 28)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Groups:
- Acthar 80U: 80 units (U) of Acthar administered 2 times a week
Arm/Group | Acthar 40U | Acthar 80U | Combined Placebo
Number analyzed (Participants) | 4 | 35 | 21
Participants | 1 | 4 | 2

ADVERSE EVENTS:
Time Frame: Week 24 plus 30 days
Description: Safety population included all randomized participants who received ≥ 1 dose of study medication.
Arm/Group | Acthar 40U | Acthar 80U | Combined Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/35 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/4 | 7/35 | 3/21
Other Adverse Events (participants affected / at risk) | 4/4 | 31/35 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar 40U (N=4) | Acthar 80U (N=35) | Combined Placebo (N=21)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acthar 40U (N=4) | Acthar 80U (N=35) | Combined Placebo (N=21)
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 5
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 0
Respiratory infection (Infections and infestations) | 0 | 0 | 2
Edema peripheral (General disorders) | 0 | 11 | 4
Fatigue (General disorders) | 1 | 2 | 2
Asthenia (General disorders) | 0 | 2 | 0
Edema (General disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 5 | 2
Nausea (Gastrointestinal disorders) | 0 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 0
Feces discolored (Gastrointestinal disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 1
Headache (Nervous system disorders) | 0 | 3 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 2
Weight increased (Investigations) | 0 | 1 | 3
Neutrophil count increased (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 5 | 0
Mood swings (Psychiatric disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Amemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator shall not, without Sponsor's prior written consent, independently publish or otherwise disclose any results of the study until a Multi-Center Publication is published. If a Multi-Center Publication is not submitted for publication within the specified timeframe, Institution and Principal Investigator shall have the right to publish and present the results of Institution's and Principal Investigator's activities solely in accordance with the Sponsor's written provisions.